CLINICAL TRIAL: NCT02008123
Title: Effect of Primidone on Platelet Responsiveness in Patients Determined to be Clopidogrel Resistant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion/Exclusion criteria was too stringent to enroll patients at this site.
Sponsor: Dent Neuroscience Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 434350-2
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Clopidogrel Resistance; Secondary Stroke Prevention
Keywords: Clopidogrel; Clopidogrel Resistance; Primidone; Secondary Stroke Prevention
MeSH Terms: interventions — Primidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primidone (Experimental): Participants will receive primidone in addition to their clopidogrel regimen. For the first 3 days of the study, participants will take 125 mg of primidone (one-half tablet). After 3 days of 125 mg, the primidone dose will be increased to 250 mg (1 tablet) taken at bedtime for the next 17-25 days. The participant will then be asked to return and be retested.
  Interventions: Drug: Primidone

INTERVENTIONS:
Drug: Primidone — Primidone is an antiepileptic used for the management of generalized tonic-clonic seizures and for the management of complex partial seizures. One of primidone's active metabolite is phenobarbital, which is a potent cytochrome P450 inducer. In this study, primidone will be used to induce CYP 1A2 in order to provide more efficient metabolism of clopidogrel to its active form
  Other Names: Mysoline (brand)

SUMMARY:
The purpose of this study is to determine whether adding primidone will improve the metabolism of clopidogrel thereby increasing metabolite levels within the blood stream and platelet response to clopidogrel in patients who were previously found to lack adequate response to clopidogrel. This information could help overcome clopidogrel resistance in patients who are at risk for stroke or transient ischemic attack (TIA).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 - 90 years who are clopidogrel resistant as determined by whole blood aggregometry
* Patients with a low risk of new cerebrovascular ischemic events as indicated by an Essen Stroke Risk Score of less than three

Exclusion Criteria:

* Any history of allergy or intolerance to either Plavix or clopidogrel
* Any history of allergy or intolerance to either Mysoline or primidone
* Any clinically significant abnormalities in complete blood count as determined by the investigator
* Use of any acute medications within the last two weeks or initiation of any non-study medications during the study period that would effect CYP enzymes or platelet function
* Use of tobacco products from 2 weeks prior to enrollment in the study and throughout the duration of the study
* Any planned surgical procedures during the study or 5 days after the study has ended
* History of alcoholism or alcohol abuse
* Participants who have had any alcohol consumption within 24 hours of a blood draw
* Previous stroke in past 3 months
* Participants who are or are planning to become pregnant
* Participants who of reproductive potential must agree to use a method of contraception for the duration of the study as well as 4 weeks after participation is complete
* Change in any medications that could affect liver enzymes or platelet aggregation throughout the study
* Compliance less than 80 % based on pill counts on two different study visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Platelet Aggregometry | Platelet aggregometry will be performed at Visit 1 and Visit 2 which will be 20-28 days following Visit 1.
  Platelet Aggregometry will be used to assess platelet responsiveness to clopidogrel following treatment with investigational medication. Blood will be placed in plastic cuvettes and probes will be inserted. Wires on the probes measure platelet aggregation in electrical impedance. A baseline is obtained and then adenosine diphosphate (ADP) is added to cause aggregation. Clopidogrel prevents platelet aggregation through irreversible binding of its active metabolite to the ADP receptors on the platelet surface. The change in impedance from baseline is directly proportional to the extent of platelet aggregation and is expressed in ohms of resistance.

SECONDARY OUTCOMES:
Area Under the Curve of Clopidogrel Metabolite Levels | Metabolite Levels Drawn 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours post clopidogrel dose at Visit 1 and Visit 2 which will be 20-28 days following Visit 1.
  Whole blood from the subjects will be drawn 30 minutes, 1 hour, 2 hours, 3 hours and 4 hours post clopidogrel dose. Once the blood is drawn, the metabolite will be derivatized to keep the metabolite stable in blood. Derivatization of the metabolite, involves spiking blood samples with 2-bromo-3'methoxyacetophenone contained in an acetonitrile solution. Once derivatization has been done, metabolite levels will be analyzed using liquid chromatography mass spectrometry (LCMS). Once concentration levels of the active metabolite are known, the area under the curve will be calculated under trapezoid rule (linear up, log down).

CONTACTS AND LOCATIONS:
Overall Officials: Vernice Bates, M.D., Principal Investigator — Dent Neurologic Institute
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States